CLINICAL TRIAL: NCT04545021
Title: Multilevel and Ecologically Grounded Assessments of Personality, Emotions and Self- Regulation as Determinants of Psychological and Physiological Adaptation in Latino Prostate Cancer Survivors Undergoing Stress Management Training
Brief Title: My Health Day by Day (Mi Salud Dia a Dia)
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Frank Penedo, Professor, University of Miami
Other Study IDs: 20190613; 1R01CA206456-01A1 (NIH)
Record Dates: First submitted 2020-08-28; First posted 2020-09-10 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Stress, Emotional
Keywords: Prostate Cancer Survivors; Cognitive Stress Management; Hispanic/Latino
MeSH Terms: conditions — Stress, Psychological

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Cognitive Behavioral Stress Management (CBSM) - PC Survivor: Participant receives standard cognitive behavioral stress management from the Parent study NCT03344757.
- CBSM - PC Survivor Partner: The survivor partner does not receive any intervention.
- Cultural CBSM (C-CBSM) - PC Survivor: Participant receives culturally adapted cognitive behavioral stress management from the Parent study NCT03344757.
- Cultural CBSM (C-CBSM) - PC Survivor Partner: The survivor partner does not receive any intervention.

SUMMARY:
The purpose of this study is to is to evaluate how Cognitive Behavioral Stress Management (CBSM) targets (e.g., anxiety reduction, cognitive reappraisal, coping, emotional expression, communication skills, social support) operate through Science of Behavior Change (SOBC) measures and influence dyadic adjustment and Health Related Quality of Life (HRQoL) in Prostate Cancer (PC) survivors and spouses/partners, in addition to physiologic adaptation and symptom burden in PC survivors.

ELIGIBILITY:
Inclusion Criteria:

Prostate Cancer Survivor

1. ≥18 years of age
2. Hispanic/Latino self- identification
3. Spanish speakers (including bilinguals who agree to participate in a Spanish intervention)
4. primary diagnosis of localized PC (T1-T3, N0, M0)
5. surgical or radiation treatment in the past 4-months
6. no history of non-skin cancer for the past 2 years
7. no psychiatric treatment or overt signs of severe psychopathology (e.g., psychosis, substance dependence)
8. owning a smartphone device with an Android or iPhone Operating System (iOS), which is necessary to collect the proposed Ecological Momentary Assessment (EMA) data or a valid email address.

(I) willingness to wear the E4 wristband at 5 time points, over the course of 4 days (J) has a spouse/partner that is willing to participate or is willing to participate in the study alone

Spouses/Partners:

1. female or male ≥18 years of age
2. have no history of inpatient psychiatric treatment for severe mental illness or overt signs of severe psychopathology (e.g., psychosis, substance dep., dementia)
3. willingness to be assessed and followed for 6 months
4. no life-threatening illness with a life expectancy < 12 months
5. identifies as a spouse/partner and is willing to participate in the study.

Exclusion Criteria:

* Not meeting all of the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The participants concurrently enrolled in the parent study NCT03344757.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-08-01 (Actual)

PRIMARY OUTCOMES:
Change in emotion regulation | Baseline to month 4, baseline to month 6
  Change in emotion regulation will be measured using the Emotion Regulation Questionnaire (ERQ). ERQ is a 10-item questionnaire with a total score ranging from 0-70 with the higher score indicating greater use of emotional regulation strategy.
Change in self regulation | Baseline to month 4, baseline to month 6
  Change in self-regulation will be measured using the Short Self-Regulation Questionnaire (SSRQ). The SSRQ is a 31-item self-report questionnaire with a total score ranging from 30-150 with the higher score indicating greater self-regulation.
Change in mindfulness attention awareness | Baseline to month 4, baseline to month 6
  Change in mindfulness attention awareness is measured using the Mindfulness Attention Awareness Scale (MAAS). MAAS has 15 questions with a total score ranging from 15-90 with the higher score indicating higher levels of dispositional mindfulness
Change in couple coercion | Baseline to month 4, baseline to month 6
  Change in couple coercion is measured using the Couple Coercion Questionnaire (CCQ). The CCQ is a 12 item questionnaire with the total score ranging from 12-72, with the higher score indicating increased perception of how coercion exemplifies his/her relationship with his/her partner.
Change in behavioral inhibition | Baseline to month 4, baseline to month 6
  Behavioral Inhibition is measured using the Behavioral Inhibition and Activation Scale (BIS/BAS). BIS/BAS scale is a 24-item questionnaire with the BIS composing of items 2, 8, 13, 16, 19, 22 and 24. The total score for BIS has a range of 7-28 with the higher score indicating increase avoidance of aversive outcomes.
Change in behavioral activation | Baseline to month 4, baseline to month 6
  Behavioral Activation is measured using the Behavioral Inhibition and Activation Scale (BIS/BAS). BIS/BAS scale is a 24-item questionnaire with the BAS composing of a subset of questions with a total score ranging from of 13-52 with the higher score indicating increased motivation to approach goal-oriented outcomes.
Change in relationship satisfaction | Baseline to month 4, baseline to month 6
  Changes in relationship satisfaction as assessed by the Revised Dyadic Adjustment Scale (RDAS). RDAS is a 14-item measure with total scores ranging from 0-69 with the higher scores indicate greater relationship satisfaction.
Heart rate variability | Up to Month 6
  Heart rate variability collected via the Empatica wrist watch
Electrodermal activity | Up to Month 6
  Electrodermal activity collected via the Empatica wrist watch
Life satisfaction as measured by the Affective Balance Scale (ABS) | Up to Month 6
  ABS is 10 item questionnaire with a total score ranging from 0-5, with the higher score indicating higher life satisfaction.
Measure of Current Status (MOCS) | Up to Month 6
  The MOCS questionnaire has a total score ranging from 0-52 with the higher score indicating increased likelihood of having the ability to relax at will.
Level of stress | Up to Month 6
  Level of stress will be measured using a Likert Scale question ranging from 1-4 with the higher value indicating greater stress.
Frequency of Text messages | Month 6
  The frequency of text messages will be reported as total amount of text messages sent and received per month, collected via Short Messaging Service (SMS) extraction software.
Length of Text messages | Month 6
  The length of text messages will be reported as average number of lines per text message collected via SMS extraction software

CONTACTS AND LOCATIONS:
Overall Officials: Frank Penedo, Ph.D., Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No